CLINICAL TRIAL: NCT02420535
Title: An Innovative Caregiver Tool to Assess and Manage Behavioral Symptoms of Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Helen Kales, Professor of Psychiatry, Director, The Program for Positive Aging Research, Associate Director for Mental Health and Aging Research,The Geriatrics Center, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: HUM00066639
Record Dates: First submitted 2015-04-14; First posted 2015-04-20 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-12

CONDITIONS: Dementia
Keywords: Dementia; Alzheimer's Disease; Caregivers; Behavioral; Caregiver burden
MeSH Terms: conditions — Dementia; Alzheimer Disease; Behavior; Caregiver Burden

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediately Receive Tool (Experimental): Caregiver/Care Recipient Dyad will be randomly assigned to immediately receive the WeCareAdvisor Tool for 4 weeks.
  Interventions: Behavioral: Immediately Receive Tool
- One Month Delay (Active Comparator): Caregiver/Care Recipient Dyad will be randomly assigned to a 4 week delay (usual care activities only) before receiving the WeCareAdvisor Tool for 4 weeks.
  Interventions: Behavioral: One Month Delay

INTERVENTIONS:
Behavioral: Immediately Receive Tool
  Arms: Immediately Receive Tool
Behavioral: One Month Delay
  Arms: One Month Delay

SUMMARY:
Behavioral symptoms that commonly occur with dementia are associated with increased health care utilization and can lead to challenges for the person living with dementia and their caregivers. Caregivers need knowledge and skills to monitor these behaviors, to identify what triggers them, and to learn how to use proven, practical medication-free strategies to prevent and manage the behaviors. The purpose of this study is to develop and test the WeCareAdvisor, a customized, internet-based computer tool for family caregivers that helps them to assess, manage and track behavioral symptoms and their contributing factors (e.g., pain, sleep disturbance), and that provides tailored strategies for in-home, medication-free behavior management. This study is a collaboration between researchers at the University of Michigan and Johns Hopkins University.

ELIGIBILITY:
Inclusion Criteria:

General

* Age 21 years or older
* Ability to read, speak and understand English
* Home location within 50 miles of the study site Caregivers (CG)
* Active primary caregiver of a Person with Dementia (PwD) for at least 6 months and planning to remain the primary caregiver for the next 2 months
* Currently living with the PwD
* CG plans to live in the area for the duration of the study
* Is familiar and comfortable utilizing technology (e.g. computers, tablets, the internet)

Persons with Dementia (PwD)

* CG reports that the PwD exhibits at least one or more behavioral symptoms (any behavior at any frequency)
* PwD receiving psychotropic medication or cognitive enhancers will not be excluded.
* If PwD is on any of four classes of psychotropic medications (antidepressant, benzodiazepines, antipsychotic, or anti-convulsant) or an anti-dementia medication (memantine or a cholinesterase inhibitor), we will require that he/she have been on a stable dose for 60 days prior to enrollment (typical time frame in clinical trials) to minimize possible confounding effects of concomitant medications.
* Clinical diagnosis of dementia (any type) or a score of less than 24 on the Mini-Mental State Examination (MMSE)

Exclusion Criteria:

General

* Inability to read, speak or understand English
* Home location greater than 50 miles from the study site
* Lack of regular access to a telephone Caregivers (CG)
* Reading literacy of less than 6th grade
* Visual impairment to the extent of prohibiting interaction with the tool
* Hearing impairment sufficient to prohibit telephone communication
* Other self-identified mental or physical health issues that would distinctly interfere with the ability to reasonably test the tool or complete behavioral interventions (e.g. substance use disorder, schizophrenia, severe mobility issues)
* Hospitalized more than 3 times in the past year
* Participating in another study to help caregivers care for the person with dementia.

Persons with Dementia (PwD)

* At a terminal phase of illness, unable to respond to the environment or with a life expectancy less than 6 months
* Active suicide risk
* Imminent placement to nursing home (within the next 60 days)
* Hospitalized more than 3 times in the past year
* Currently in another study testing a medication to control behavioral symptoms

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2015-05; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Effects of the WeCareAdvisor Tool on Caregiver Upset | 4 weeks
  We will measure caregiver upset on a 5 point rating scale "not at all", "a little", "moderately", "very much" and "extremely"
Effect of the WeCareAdvisor Tool on Caregiver Confidence | 4 weeks
  We will measure caregiver confidence on a 5 point rating scale "not at all", "a little", "moderately", "very much" and "extremely"

CONTACTS AND LOCATIONS:
Overall Officials: Helen Kales, MD, Principal Investigator — University of Michigan; Laura Gitlin, PhD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins School of Nursing, Baltimore, Maryland
  - University of Michigan Department of Psychiatry, Ann Arbor, Michigan

REFERENCES:
- [Derived] Gonzalez-Fraile E, Ballesteros J, Rueda JR, Santos-Zorrozua B, Sola I, McCleery J. Remotely delivered information, training and support for informal caregivers of people with dementia. Cochrane Database Syst Rev. 2021 Jan 4;1(1):CD006440. doi: 10.1002/14651858.CD006440.pub3. PMID 33417236
- [Derived] Kales HC, Gitlin LN, Stanislawski B, Myra Kim H, Marx K, Turnwald M, Chiang C, Lyketsos CG. Effect of the WeCareAdvisor on family caregiver outcomes in dementia: a pilot randomized controlled trial. BMC Geriatr. 2018 May 10;18(1):113. doi: 10.1186/s12877-018-0801-8. PMID 29747583
- [Derived] Gitlin LN, Kales HC, Marx K, Stanislawski B, Lyketsos C. A randomized trial of a web-based platform to help families manage dementia-related behavioral symptoms: The WeCareAdvisor. Contemp Clin Trials. 2017 Nov;62:27-36. doi: 10.1016/j.cct.2017.08.001. Epub 2017 Aug 9. PMID 28800895